CLINICAL TRIAL: NCT03039959
Title: Predictive Value of Renal Venous Flow Profiles for Adverse Outcomes in Right Heart Failure
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Faeq Husain, Senior Physician Nephrology, University of Giessen
Other Study IDs: AZ 237/16
Record Dates: First submitted 2017-01-29; First posted 2017-02-01 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Pulmonary Hypertension; Cardiorenal Syndrome; Heart Failure
Keywords: Renal Doppler ultrasonography; Venous Congestion
MeSH Terms: conditions — Hypertension, Pulmonary; Cardio-Renal Syndrome; Heart Failure; Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — Only residual material will be reserved for the Deutsche Zentrum für Lungenforschung Biobank
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulmonary hypertension cohort: Consecutive adult Pulmonology inpatients with suspected or pre-diagnosed pulmonary hypertension undergoing invasive right heart catheterization.
  Interventions: Diagnostic Test: No intervention
- Heart failure cohort: Consecutive adult Cardiology inpatients with a new or pre-existing diagnosis of heart failure who are referred to the consultant nephrologist with a history of diuretic-resistant fluid overload and impaired renal function.
  Interventions: Diagnostic Test: No intervention

INTERVENTIONS:
Diagnostic Test: No intervention — No intervention

SUMMARY:
Predictive value of renal venous flow profiles for adverse outcomes in patients with right heart failure

DETAILED DESCRIPTION:
Persistent congestion with deteriorating renal function is an important cause of adverse outcomes in heart failure. The investigators aimed to characterize new Doppler ultrasonography approaches to evaluate the continuum of renal congestion. Pulmonary hypertension is the most common precursor to right heart failure and thus represents an ideal scenario to study congestion. The second cohort comprises consecutive Cardiology inpatients aged ≥18 years with a new or pre-existing diagnosis of heart failure who are referred to the consultant nephrologist with a history of diuretic-resistant fluid overload and impaired renal function. The investigators choose patients with heart failure to broaden the findings to the most common clinical entity of right ventricular failure.

ELIGIBILITY:
Pulmonary hypertension cohort:

Exclusion Criteria:

* CKD stage 5 (KDIGO)
* pre-existing acute kidney injury (acute kidney injury was defined as an increase in serum creatinine by ≥ 0.3 mg/dl within 48 hours or to ≥ 1.5 times baseline within the prior 7 days, as determined by all available serum creatinine values from hospital and outpatient medical records within the previous 90 days)
* Non-end stage renal disease patients with extracorporeal or peritoneal ultrafiltration for treatment of diuretic-resistant fluid overload
* Patients with primary kidney disease (e.g., glomerulonephritis, autosomal dominant polycystic kidney disease, postrenal obstruction)
* solid-organ transplant recipients
* use of non-steroidal inflammatory drugs within 72 hours before right heart catheterization

Heart failure cohort:

Exclusion criteria same as in the discovery cohort except pre-existing acute kidney injury

* Patients with mechanical assist devices are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive Pulmonology inpatients with suspected or pre-diagnosed pulmonary hypertension undergoing right heart catheterization (pulmonary hypertension cohort) and consecutive Cardiology inpatients who are referred to the consultant nephrologist with a history of diuretic-resistant fluid overload and impaired renal function (heart failure cohort).
Sampling Method: Probability Sample
Enrollment: 421 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Rate of pulmonary hypertension-related morbidity and all-cause mortality (pulmonary hypertension cohort) | 1 year post-discharge
  Any hospitalization for worsening of pulmonary hypertension, lung transplantation, or need for escalation of pulmonary hypertension-specific therapy, and death from any cause
First occurrence of worsening heart failure and first occurrence of need for renal replacement therapy (heart failure cohort) | 1 year post-discharge
  Unscheduled hospitalization or unscheduled office visit for heart failure and new onset renal replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: Werner Seeger, MD, Study Director — Department of Internal Medicine II; Division of Pulmonology, Nephrology and Critical Care Medicine
Locations (1):
- University Clinic Giessen and Marburg - Campus Giessen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Navaneethan SD, Wehbe E, Heresi GA, Gaur V, Minai OA, Arrigain S, Nally JV Jr, Schold JD, Rahman M, Dweik RA. Presence and outcomes of kidney disease in patients with pulmonary hypertension. Clin J Am Soc Nephrol. 2014 May;9(5):855-63. doi: 10.2215/CJN.10191013. Epub 2014 Feb 27. PMID 24578332
- [Result] Iida N, Seo Y, Sai S, Machino-Ohtsuka T, Yamamoto M, Ishizu T, Kawakami Y, Aonuma K. Clinical Implications of Intrarenal Hemodynamic Evaluation by Doppler Ultrasonography in Heart Failure. JACC Heart Fail. 2016 Aug;4(8):674-82. doi: 10.1016/j.jchf.2016.03.016. Epub 2016 May 11. PMID 27179835
- [Result] Sugiura T, Wada A. Resistive index predicts renal prognosis in chronic kidney disease. Nephrol Dial Transplant. 2009 Sep;24(9):2780-5. doi: 10.1093/ndt/gfp121. Epub 2009 Mar 23. PMID 19318356
- [Derived] Kuhnert S, Sommerlad J, Gall H, Weder MM, Wolff M, Eberle S, Sander M, Reichert M, Koch C, Askevold I, Hecker A, Padberg W, Ostermann M, Mehta R, Ronco C, Birk HW, Seeger W, Mayer K, Hecker M, Husain-Syed F. Postoperative Fluid Accumulation is Associated With Underestimation of AKI Severity in Lung Transplant Recipients. Clin Transplant. 2024 Sep;38(9):e15457. doi: 10.1111/ctr.15457. PMID 39282762
- [Derived] Husain-Syed F, Singam NSV, Viehman JK, Vaughan L, Bauer P, Gall H, Tello K, Richter MJ, Yogeswaran A, Romero-Gonzalez G, Rosner MH, Ronco C, Assmus B, Ghofrani HA, Seeger W, Birk HW, Kashani KB. Changes in Doppler-Derived Kidney Venous Flow and Adverse Cardiorenal Outcomes in Patients With Heart Failure. J Am Heart Assoc. 2023 Aug 15;12(16):e030145. doi: 10.1161/JAHA.123.030145. Epub 2023 Aug 14. PMID 37577933
- [Derived] Husain-Syed F, Birk HW, Ronco C, Schormann T, Tello K, Richter MJ, Wilhelm J, Sommer N, Steyerberg E, Bauer P, Walmrath HD, Seeger W, McCullough PA, Gall H, Ghofrani HA. Doppler-Derived Renal Venous Stasis Index in the Prognosis of Right Heart Failure. J Am Heart Assoc. 2019 Nov 5;8(21):e013584. doi: 10.1161/JAHA.119.013584. Epub 2019 Oct 19. PMID 31630601